CLINICAL TRIAL: NCT03144687
Title: An Open-Label Phase 2 Study of Itacitinib (INCB039110) in Combination With Low-Dose Ruxolitinib or Itacitinib Alone Following Ruxolitinib in Subjects With Myelofibrosis
Brief Title: A Study of Itacitinib in Combination With Low-Dose Ruxolitinib or Itacitinib Alone Following Ruxolitinib in Participants With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-209; 2017-005109-11 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Myelofibrosis; Janus kinase (JAK) inhibitor; itacitinib; ruxolitinib
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis | interventions — itacitinib; INCB039110; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants with MF who were tolerating a ruxolitinib dose of less than 20 milligrams (mg) daily with no dose increase or no dose modification in the 8 weeks before screening visit received a combination of the itacitinib at the dose of 200 mg, orally, once daily (QD) and ruxolitinib, orally, twice daily (BID) at their previous stable dose (must had been < 20 mg daily). Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment are met.
  Interventions: Drug: Itacitinib; Drug: Ruxolitinib
- Cohort B (Experimental): Participants with MF who progressed after initial reduction in spleen with ruxolitinib treatment, progressed or discontinued for hematologic toxicities received treatment with itacitinib alone at the dose of 600 mg QD. Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment are met.
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — Itacitinib self-administered orally once daily .
  Other Names: INCB039110
Drug: Ruxolitinib — Ruxolitinib self-administered orally at the stable dose of < 20 mg daily established before entering the study.
  Other Names: INCB018424; Jakafi; Jakavi
  Arms: Cohort A

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of itacitinib combined with low-dose ruxolitinib or itacitinib alone in participants with myelofibrosis (MF).

ELIGIBILITY:
Inclusion Criteria:

Cohort A only

•Receiving ruxolitinib dose of less than 20 mg daily with no dose increase or no dose modification in the last 8 weeks before screening visit.

Cohort B only

•Must have had initial reduction in spleen on ruxolitinib treatment:

* Followed by documented evidence of progression in spleen length or volume OR
* Discontinued ruxolitinib for hematologic toxicities, after the initial reduction in spleen length or volume.

All participants

* Confirmed diagnosis of primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis according to revised World Health Organization 2016 criteria.
* Must have palpable spleen of greater than or equal to (≥) 5 centimeter (cm) below the left subcostal margin on physical examination at the screening visit.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
* Screening bone marrow biopsy specimen available or willingness to undergo a bone marrow biopsy at screening/baseline; willingness to undergo bone marrow biopsy at Week 24.
* Life expectancy of at least 24 weeks.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Lack of recovery from all toxicities from previous therapy (except ruxolitinib) to Grade 1 or better.
* Previous treatment with itacitinib or Janus kinase (JAK1) inhibitors (JAK1/JAK2 inhibitor ruxolitinib is permitted).
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* Recent history of inadequate bone marrow reserve as demonstrated by protocol-defined criteria.
* Inadequate liver function at screening and baseline visits as demonstrated by protocol-defined criteria.
* Inadequate renal function at screening and baseline visits as demonstrated by protocol-defined criteria.
* Active bacterial, fungal, parasitic, or viral infection that requires therapy.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation: HBV deoxyribonucleic acid (DNA) and HCV ribonucleic acid (RNA) must be undetectable. Participants cannot be positive for hepatitis B surface antigen or anti-hepatitis B core antibodies. Participants who have positive anti-HBs as the only evidence of prior exposure may participate in the study provided that there is both 1) no known history of HBV infection and 2) verified receipt of hepatitis B vaccine.
* Known human immunodeficiency virus infection.
* Clinically significant or uncontrolled cardiac disease.
* Active invasive malignancy over the previous 2 years except treated basal or squamous carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, and completely resected papillary thyroid and follicular thyroid cancers. Participants with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery may be enrolled as long as they have a reasonable expectation to have been cured with the treatment modality received.
* Splenic irradiation within 6 months before receiving the first dose of itacitinib.
* Use of any prohibited concomitant medications.
* Active alcohol or drug addiction that would interfere with their ability to comply with the study requirements.
* Use of any potent/strong cytochrome P450 3A4 inhibitors within 14 days or 5 half-lives (whichever is longer) before the first dose of itacitinib or anticipated during the study.
* Use of concomitant treatment of fluconazole at a dose > 200 mg (for ruxolitinib participants treated in Cohort A only).
* Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
* Currently breastfeeding or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, Study Director — Incyte Corporation
Locations (26):
- United States (19):
  - Arizona Oncology Associates, Tempe, Arizona
  - UC Irvine Medical Center, Orange, California
  - Anschutz Cancer Pavilion - University Of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Nebraska Cancer Specialist, Omaha, Nebraska
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Willamette Valley Cancer Institute, Eugene, Oregon
  - Consultants in Medical Oncology and Hematology, PC, Broomall, Pennsylvania
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
- Austria (3):
  - Ordensklinikum Linz GmbH, Servicestelle für Studien, Linz
  - Paracelsus Medical University Salzburg, Salzburg
  - Hanusch Hospital, Vienna
- Netherlands (4):
  - VU Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht Department of Hematology, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 study centers in the United States, 1 study center in Austria, and 1 study center in the Netherlands.
Pre-assignment Details: A total of 23 participants with Myelofibrosis (MF) were enrolled in the study and received itacitinib + ruxolitinib (Cohort A) or itacitinib monotherapy (Cohort B).
Groups:
- Cohort A: Participants with MF who were tolerating a ruxolitinib dose of less than 20 milligrams (mg) daily with no dose increase or no dose modification in the 8 weeks before screening visit received a combination of itacitinib at the dose of 200 mg, orally, once daily (QD) and ruxolitinib, orally, twice daily (BID) at their previous stable dose (must had been < 20 mg daily). Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment were met.
- Cohort B: Participants with MF who progressed after initial reduction in spleen with ruxolitinib treatment, progressed or discontinued for hematologic toxicities received treatment with itacitinib alone at the dose of 600 mg QD. Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment were met.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 13 | 10
Completed | 10 | 3
Not Completed | 3 | 7
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Not Reported | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (6.20) | 72.0 (7.33) | 70.8 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 9 | 21
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 13 | 8 | 21
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Spleen Volume at Week 24 Compared to Baseline
Description: Spleen volume was measured using magnetic resonance imaging (MRI) or CT scan in participants who were not candidates for MRI or when MRI was not readily available. The MRIs or CTs were read in the central imaging laboratory. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the technique of least squares. The same method (MRI or CT) was used for a given participant unless a new contraindication to the use of MRI (eg, pacemaker insertion) occurred. A positive value indicates an increase in spleen volume and a negative value indicates a decrease in spleen volume.
Time Frame: Baseline and Week 24
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib. Here, Overall Number of participants analyzed ("N") signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 5
cubic centimeter (cm^3) | 88.7 (563.5) | -207 (571.3)

2. Primary Outcome: Percentage Change in Spleen Volume at Week 24 Compared to Baseline
Description: Spleen volume was measured using MRI or CT scan in participants who were not candidates for MRI or when MRI was not readily available. The MRIs or CTs were read in the central imaging laboratory. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the technique of least squares. The same method (MRI or CT) was used for a given participant unless a new contraindication to the use of MRI (eg, pacemaker insertion) occurred. A positive value indicates an increase in spleen volume and a negative value indicates a decrease in spleen volume.
Time Frame: Baseline and Week 24
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib. Here, "N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 5
percentage change | 6.9 (27.49) | -3.0 (34.67)

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether considered drug related, that occurs after a participant provides informed consent. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug. An SAE is an AE resulting in: death; initial/prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly.
Time Frame: up to approximately 40 months (3.3 years)
Population: Safety Population included all enrolled participants who received at least 1 dose of itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 13 | 10
Participants
  TEAE | 13 | 10
  SAE | 3 | 5

4. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology, clinical chemistry, coagulation and urinalysis. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Time Frame: up to approximately 40 months (3.3 years)
Population: Safety Population included all enrolled participants who received at least 1 dose of itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 13 | 10
Participants
  Hemoglobin: High Direction | 0 | 0
  Hemoglobin: Low Direction | 4 | 4
  Leukocytes: High Direction | 0 | 1
  Leukocytes: Low Direction | 0 | 0
  Lymphocytes: High Direction | 0 | 0
  Lymphocytes: Low Direction | 3 | 1
  Neutrophils | 0 | 1
  Platelets | 3 | 4
  Alanine Aminotransferase | 0 | 0
  Albumin | 0 | 0
  Alkaline Phosphatase | 0 | 0
  Aspartate Aminotransferase | 0 | 0
  Bilirubin | 1 | 0
  Calcium: High Direction | 0 | 0
  Calcium: Low Direction | 0 | 0
  Cholesterol | 0 | 0
  Creatinine | 0 | 0
  Glucose: High Direction | 0 | 0
  Glucose: Low Direction | 0 | 0
  Phosphate | 0 | 1
  Potassium: High Direction | 0 | 0
  Potassium: Low Direction | 0 | 0
  Sodium: High Direction | 0 | 0
  Sodium: Low Direction | 0 | 0
  Triglycerides | 0 | 1
  Urate | 1 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure, pulse rate, respiratory rate, weight and height. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in vital signs were reported.
Time Frame: up to approximately 40 months (3.3 years)
Population: Safety Population included all enrolled participants who received at least 1 dose of itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 13 | 10
Participants
  Systolic blood pressure, Week 12 | 1 | 1
  Systolic blood pressure, Week 24 | 0 | 1
  Systolic blood pressure, Week 36 | 0 | 1
  Systolic blood pressure, End of Treatment | 1 | 0
  Diastolic blood pressure, Week 12 | 0 | 1
  Pulse, Week 84 | 1 | 0
  Pulse, Follow-up | 1 | 0

6. Secondary Outcome: Change From Baseline Through Week 12 in SVR as Measured by MRI (or CT Scan in Applicable Participants)
Description: Spleen volume was measured using magnetic resonance imaging (or CT scan in applicable participants). MRI of the upper and lower abdomen and pelvis was performed, to assess spleen volumes. MRI was performed with a body coil. The MRIs were read in the central imaging laboratory. Spleen volume was obtained by outlining the circumference of the organ and determining the volume using the technique of least squares. MRI was the preferred method for obtaining spleen volume data. The CT scans were processed by the same central laboratory used for MRIs. The same method (MRI or CT) was used for a given participant unless a new contraindication to the use of MRI (eg, pacemaker insertion) occurred.
Time Frame: Baseline through Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 8
cm^3 | -29.2 (349.3) | -608 (669.6)

7. Secondary Outcome: Percentage Change From Baseline Through Week 12 in SVR as Measured by MRI (or CT Scan in Applicable Participants)
Description: as for outcome 6
Time Frame: Baseline through Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 8
percentage change | -1.6 (14.69) | -24.6 (21.72)

8. Secondary Outcome: Change From Baseline Through Week 12 and Week 24 on Spleen Length as Measured by Palpation
Description: Measurement of spleen length below the left costal margin was measured by palpation. Spleen size was determined at every physical examination with the participant in the recumbent (not left decubitus) position. The edge of the spleen was determined by palpation, and measured in centimeters, using a soft ruler, from the costal margin to the point of greatest splenic protrusion. The measurements should be noted and the site at which it was determined listed (eg, anterior axillary line, midclavicular line, and/or subxiphoid). A positive value indicates an increase in spleen volume and a negative value indicates a decrease in spleen volume.
Time Frame: Baseline through Weeks 12 and 24
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib. Here, "N "signifies number of participants analyzed for this outcome measure and "n" signifies number of participants with data available at a particular time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 7
cm
  Week 12 | -0.2 (2.17) | -3.6 (6.73)
  Week 24: number analyzed (Participants) | 9 | 5
  Week 24 | -0.4 (5.41) | -2.6 (3.44)

9. Secondary Outcome: Percentage Change From Baseline Through Week 12 and Week 24 on Spleen Length as Measured by Palpation
Description: as for outcome 8
Time Frame: Baseline through Weeks 12 and 24
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib. Here, "N" signifies number of participants analyzed for this outcome measure and "n" signifies number of participants with data available at a particular time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 7
percentage change
  Week 12 | 8.8 (40.83) | -14.4 (49.89)
  Week 24: number analyzed (Participants) | 9 | 5
  Week 24 | 2.5 (50.72) | -21.3 (27.94)

10. Secondary Outcome: Change From Baseline Through Week 12 and Week 24 in Total Symptom Score as Measured by the Myelofibrosis Symptom Assessment Form (MFSAF) v2.0 Symptom Diary
Description: Symptoms of myelofibrosis were assessed using a modified MFSAF Version 2.0 diary. Using the diary, participants rated the following symptoms on a scale from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be): itching, night sweats, abdominal discomfort/bloating, early satiety, pain under the ribs on left side and bone/muscle pain. The total symptom score ranged from 0-60 and was calculated as the sum of the 6 symptom scores. A higher score indicates worse symptoms.
Time Frame: Baseline through Weeks 12 and 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 7
score on scale
  Change at Week 12 | 1.4 (6.06) | -4.7 (12.50)
  Change at Week 24: number analyzed (Participants) | 9 | 5
  Change at Week 24 | -1.0 (9.88) | -0.3 (10.14)

11. Secondary Outcome: Percentage Change From Baseline Through Week 12 and Week 24 in Total Symptom Score as Measured by the MFSAF v2.0 Symptom Diary
Description: as for outcome 10
Time Frame: Baseline through Weeks 12 and 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 6
percentage change
  Percentage Change at Week 12 | 0.7 (69.57) | -1.8 (116.6)
  Percentage Change at Week 24: number analyzed (Participants) | 9 | 4
  Percentage Change at Week 24 | -5.6 (95.56) | 33.7 (142.3)

12. Secondary Outcome: Change From Baseline Through Week 12 and Week 24 in Total Symptom Score as Measured by the Myeloproliferative Neoplasm-Symptom Assessment Form (MPN-SAF)
Description: Symptoms are evaluated by the MPN-SAF TSS. The MPN-SAF TSS assessed by the participants themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). A higher score indicates worse symptoms.
Time Frame: Baseline through Week 12 and Week 24
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib. . Here, "N" signifies number of participants analyzed for this outcome measure and "n" signifies number of participants with data available at a particular time point.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 7
score on scale
  Change at Week 12 | 2.0 (9.76) | -3.7 (12.91)
  Change at Week 24: number analyzed (Participants) | 9 | 4
  Change at Week 24 | -1.6 (11.11) | -6.0 (8.76)

13. Secondary Outcome: Percentage Change From Baseline Through Week 12 and Week 24 in Total Symptom Score as Measured by the MPN-SAF
Description: Symptoms are evaluated by the MPN-SAF TSS. The MPN-SAF TSS assessed by the participants themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). A higher score indicates worse symptoms. Note that the mean percentage change can vary in direction from the mean absolute change because percent increases (but not decreases) can exceed 100%.
Time Frame: Baseline through Week 12 and Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 7
percentage change
  Percentage Change at Week 12 | 3.8 (47.25) | -6.1 (51.24)
  Percentage Change at Week 24: number analyzed (Participants) | 9 | 4
  Percentage Change at Week 24 | 5.8 (46.85) | -22.7 (29.62)

14. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Each Visit
Description: Symptoms of myelofibrosis were assessed using the PGIC questionnaire. Using the questionnaire, participants rated the overall sense of treatment effect on their symptoms on a scale of 1 (very much improved)- 7(very much worse). The specific wording was: Since the start of the treatment you have received in this study, your myelofibrosis symptoms are: 1) Very much improved, 2) Much improved, 3) Minimally improved, 4) No change, 5) Minimally worse, 6) Much worse, 7) Very much worse. A higher score indicates worse symptoms.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, and 168
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 11 | 9
score on scale
  Week 4: number analyzed (Participants) | 11 | 8
  Week 4 | 3.6 (0.81) | 3.5 (0.93)
  Weeks 8 | 3.3 (0.90) | 3.3 (1.22)
  Weeks 12: number analyzed (Participants) | 11 | 7
  Weeks 12 | 3.2 (0.98) | 3.6 (0.98)
  Weeks 16: number analyzed (Participants) | 9 | 6
  Weeks 16 | 3.0 (1.00) | 4.2 (1.47)
  Weeks 20: number analyzed (Participants) | 8 | 6
  Weeks 20 | 3.3 (0.71) | 3.2 (0.75)
  Weeks 24: number analyzed (Participants) | 9 | 4
  Weeks 24 | 3.2 (1.09) | 2.8 (0.96)
  Weeks 36: number analyzed (Participants) | 6 | 3
  Weeks 36 | 3.2 (0.98) | 3.0 (1.00)
  Weeks 48: number analyzed (Participants) | 4 | 1
  Weeks 48 | 2.5 (1.00) | 2.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Weeks 60: number analyzed (Participants) | 3 | 1
  Weeks 60 | 3.0 (1.73) | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Weeks 72: number analyzed (Participants) | 4 | 1
  Weeks 72 | 3.3 (1.50) | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Weeks 84: number analyzed (Participants) | 1 | 1
  Weeks 84 | 2.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Weeks 96: number analyzed (Participants) | 0 | 1
  Weeks 96 |  | 2.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Weeks 108: number analyzed (Participants) | 0 | 1
  Weeks 108 |  | 4.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 120: number analyzed (Participants) | 0 | 1
  Week 120 |  | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 132: number analyzed (Participants) | 0 | 1
  Week 132 |  | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 168: number analyzed (Participants) | 0 | 1
  Week 168 |  | 3.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

15. Secondary Outcome: Number of Participants With Responses According to the 2013 International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Consensus Criteria for Treatment Response
Description: Treatment response (complete remission [CR] or partial remission [PR]) graded per IWG-MRT. CR: Bone marrow (BM): < 5% blasts; ≤ Grade 1 MF, Peripheral blood: Hemoglobin (Hb) ≥ 100 grams per liter (g/L), < upper normal limit (UNL); neutrophil count ≥ 1 × 10^9/L and < UNL; Platelet count ≥ 100 × 10^9/L and < UNL; < 2% immature myeloid cells (IMCs) and Clinical: Resolution of disease symptoms; spleen, liver not palpable; no evidence of extramedullary hematopoeisis (EMH). PR: Peripheral blood: Hb ≥ 100 g/L and < UNL; neutrophil count ≥ 1 × 10^9/L and < UNL; platelet count ≥ 100 × 10^9/L and < UNL; < 2% IMCs and Clinical: Resolution of symptoms; spleen and liver not palpable; no evidence of EMH or BM: < 5% blasts; ≤ Grade 1 MF; and peripheral blood: Hb≥ 85 g/L but < 100 g/L and < UNL; neutrophil count ≥ 1 × 10^9/L and < UNL; platelet count ≥ 50 × 10^9/L but < 100 × 10^9/L and < UNL; < 2% IMCs and Clinical: Resolution of symptoms; spleen, liver not palpable; no evidence of EMH.
Time Frame: up to approximately 40 months (3.3 years)
Population: Full Analysis Set included all enrolled participants who received at least 1 dose of itacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

16. Secondary Outcome: Area Under the Concentration-time Curve Over a Dosing Interval (AUCtau) for Itacitinib
Description: AUCtau defined as area under the concentration-time curve over a dosing interval for Itacitinib. The concentrations of itacitinib in plasma were determined using a validated Liquid Chromatography with tandem mass spectrometry (LC/MS/MS) method with an assay range of 5 to 5000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ). Itacitinib PK data for Cohort A on Week 2 were not available as itacitinib was to be held until the completion of PK sample collection.
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: Pharmacokinetic evaluable population included all participants who received at least 1 dose of itacitinib and provided at least 1 post-dose plasma sample for PK. Here, "N " signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanomolar* hour (nM*h)
Groups:
- PK: Cohort A (Itacitinib): Participants received itacitinib at the dose of 200 mg, orally, QD. Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment are met.
- PK: Cohort B (Itacitinib): Participants itacitinib alone at the dose of 600 mg QD. Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment are met.
Arm/Group | PK: Cohort A (Itacitinib) | PK: Cohort B (Itacitinib)
Number analyzed (Participants) | 12 | 8
nanomolar* hour (nM*h)
  Week 2: number analyzed (Participants) | 0 | 8
  Week 2 |  | 24100 (6600)
  Week 4: number analyzed (Participants) | 12 | 7
  Week 4 | 2540 (2020) | 28900 (11200)

17. Secondary Outcome: Area Under the Concentration-time Curve Over a Dosing Interval (AUCtau) for Ruxolitinib
Description: AUCtau defined as area under the concentration-time curve over a dosing interval for ruxolitinib. The concentrations of ruxolitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 1 to 1000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ).
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: Pharmacokinetic evaluable population included all participants who received at least 1 dose of ruxolitinib and provided at least 1 post-dose plasma sample for PK. Here, "N " signifies number of participants analyzed for this outcome measure. Only the data from 15mg QD is shown as it is the only dose level with at least three participants at both week 2 and week 4.
Measure: Mean (Standard Deviation); unit: nM*h
Groups:
- PK: Cohort A (Ruxolitinib): Participants received ruxolitinib, orally, BID at their previous stable dose (must have been < 20 mg daily). Participants continued study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or other Protocol-specified criteria to stop treatment are met.
Arm/Group | PK: Cohort A (Ruxolitinib)
Number analyzed (Participants) | 4
nM*h
  Week 2: number analyzed (Participants) | 3
  Week 2 | 2930 (486)
  Week 4 | 2350 (635)

18. Secondary Outcome: Apparent Oral Dose Clearance (CL/F) of Itacitinib
Description: Clearance of a drug was measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The concentrations of itacitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 5 to 5000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ). Data for Cohort A (Itacitinib) on Week 2 was not available as Cohort A, itacitinib was to be held on Week 2 until the completion of the PK sample collection.
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | PK: Cohort A (Itacitinib) | PK: Cohort B (Itacitinib)
Number analyzed (Participants) | 12 | 8
liters per hour (L/h)
  Week 2: number analyzed (Participants) | 0 | 8
  Week 2 |  | 48.5 (14.9)
  Week 4: number analyzed (Participants) | 12 | 7
  Week 4 | 203 (97.4) | 42.4 (15.8)

19. Secondary Outcome: Apparent Oral Dose Clearance (CL/F) of Ruxolitinib
Description: Clearance of a drug was measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The concentrations of ruxolitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 1 to 1000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ).
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | PK: Cohort A (Ruxolitinib)
Number analyzed (Participants) | 4
L/h
  Week 2: number analyzed (Participants) | 3
  Week 2 | 17.0 (3.12)
  Week 4 | 22.2 (6.82)

20. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Itacitinib
Description: The concentrations of itacitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 5 to 5000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ). Data for Cohort A (Itacitinib) on Week 2 was not available as Cohort A, itacitinib was to be held on Week 2 until the completion of the PK sample collection.
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nanometer (nM)
Arm/Group | PK: Cohort A (Itacitinib) | PK: Cohort B (Itacitinib)
Number analyzed (Participants) | 12 | 8
nanometer (nM)
  Week 2: number analyzed (Participants) | 0 | 8
  Week 2 |  | 3570 (1280)
  Week 4: number analyzed (Participants) | 12 | 7
  Week 4 | 559 (518) | 4460 (2470)

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ruxolitinib
Description: The concentrations of ruxolitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 1 to 1000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ).
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | PK: Cohort A (Ruxolitinib)
Number analyzed (Participants) | 4
nM
  Week 2: number analyzed (Participants) | 3
  Week 2 | 695 (111)
  Week 4 | 677 (118)

22. Secondary Outcome: Time to Maximum Concentration (Tmax) of Itacitinib
Description: as for outcome 20
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 16
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PK: Cohort A (Itacitinib) | PK: Cohort B (Itacitinib)
Number analyzed (Participants) | 12 | 8
hour (hr)
  Week 2: number analyzed (Participants) | 0 | 8
  Week 2 |  | 2.0 [1.0 to 5.0]
  Week 4: number analyzed (Participants) | 12 | 7
  Week 4 | 2.0 [1.0 to 2.3] | 2.0 [2.0 to 4.6]

23. Secondary Outcome: Time to Maximum Concentration (Tmax) of Ruxolitinib
Description: as for outcome 21
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 17
Measure: Median (Full Range); unit: hr
Arm/Group | PK: Cohort A (Ruxolitinib)
Number analyzed (Participants) | 4
hr
  Week 2: number analyzed (Participants) | 3
  Week 2 | 1.0 [1.0 to 1.1]
  Week 4 | 1.0 [1.0 to 1.1]

24. Secondary Outcome: Concentration at the End of the Dosing Interval (Ctau) of Itacitinib
Description: Ctau is defined as concentration at the end of the dosing interval of ruxolitinib.The concentrations of itacitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 5 to 5000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ). Data for Cohort A (Itacitinib) on Week 2 was not available as Cohort A, itacitinib was to be held on Week 2 until the completion of the PK sample collection.
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose on Week 2 and Week 4
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | PK: Cohort A (Itacitinib) | PK: Cohort B (Itacitinib)
Number analyzed (Participants) | 12 | 9
nM
  Week 2: number analyzed (Participants) | 0 | 8
  Week 2 |  | 102 (120)
  Week 4 | 10.2 (8.67) | 108 (85.4)

25. Secondary Outcome: Concentration at the End of the Dosing Interval (Ctau) of Ruxolitinib
Description: Ctau is defined as concentration at the end of the dosing interval of ruxolitinib. The concentrations of ruxolitinib in plasma were determined using a validated LC/MS/MS method with an assay range of 1 to 1000 nM. The PK parameters were calculated using standard noncompartmental analysis in Phoenix WinNonlin® v8.2 (Certara USA Inc., Princeton, NJ).
Time Frame: 0 (pre-dose), 1, 2, 5 and 8 hours post-dose Week 2 and Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | PK: Cohort A (Ruxolitinib)
Number analyzed (Participants) | 4
nM
  Week 2: number analyzed (Participants) | 3
  Week 2 | 16.6 (14.5)
  Week 4 | 19.7 (28.6)

ADVERSE EVENTS:
Time Frame: up to approximately 40 months (3.3 years)
Groups:
- Total: Total
Arm/Group | Cohort A | Cohort B | Total
All-Cause Mortality (participants affected / at risk) | 0/13 | 2/10 | 2/23
Serious Adverse Events (participants affected / at risk) | 3/13 | 5/10 | 8/23
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=13) | Cohort B (N=10) | Total (N=23)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Stent removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=13) | Cohort B (N=10) | Total (N=23)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (10) | 8 (14)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 1 (1) | 3 (4)
Blood chloride increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 1 (2) | 2 (4)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Calcinosis (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (8) | 8 (12)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 5 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
Fatigue (General disorders) | 3 (3) | 5 (6) | 8 (9)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 3 (5)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (5) | 5 (7)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (2) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2)
Posterior tibial tendon dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 4 (6) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Reticulocyte count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 2 (2) | 4 (7)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (6) | 2 (3) | 5 (9)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03144687/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03144687/SAP_001.pdf